CLINICAL TRIAL: NCT04832360
Title: Testing Financial Incentive Interventions in Dyadic-Smoker Couples
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Responsible Party: Principal Investigator, Michelle R Vandellen, Associate Professor, Principal Investigator, University of Georgia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RCA241570A
Record Dates: First submitted 2021-01-08; First posted 2021-04-05 (Actual); Results first posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (CTL) (Experimental): Participants do not receive financial incentive intervention
  Interventions: Behavioral: Financial Incentives
- Single Target (ST) (Experimental): One member of each dyadic-smoking couple will receive financial incentive intervention
  Interventions: Behavioral: Financial Incentives
- Dyadic Target (DT) (Experimental): Both members of each dyadic-smoking couple will receive financial incentive intervention
  Interventions: Behavioral: Financial Incentives

INTERVENTIONS:
Behavioral: Financial Incentives — Financial incentives may be offered to participants based on their behavioral outcomes (smoking cessation and participation in online psychoeducation about smoking)

SUMMARY:
The proposed study investigates the feasibility and efficacy of FITs in dual-smoker couples [DSCs]. The core design is a three-group mixed repeated measures design, in which participants are randomized into one of three conditions (control [CTL], dyadic target [DT] FIT or single target [ST] FIT) and tracked across 3 months. The FIT involves monetary incentives for online psychoeducation completion and smoking abstinence at follow-up.

DETAILED DESCRIPTION:
The proposed study investigates the feasibility and efficacy of FITs in dual-smoker couples [DSCs]. The core design is a three-group mixed repeated measures design, in which participants are randomized into one of three conditions (control [CTL], dyadic target [DT] FIT or single target [ST] FIT) and tracked across 3 months. During this time, participants will complete a baseline session and a follow-up. Between these visits, all participants will have access to a voluntary brief cessation program (i.e., online psychoeducation created for this study using Beat the Pack materials and resources from NCI, NIH + Nicotine Replacement Therapy [NRT]). The FIT involves monetary incentives for online psychoeducation completion and smoking abstinence at follow-up. In the ST condition, one member of each couple (i.e., the target) will receive monetary incentives; in the DT condition, both members of the couple will receive monetary incentives. This design allows for preliminary consideration of FITs in DSCs and tests whether FITs for both members of the dyad synergistically enhances outcomes.

ELIGIBILITY:
Inclusion Criteria:

both members:

* age of 18+
* smoke 5+ combustible cigarettes/day
* may not have participated in pilot study

Exclusion Criteria:

* < 8th grade capacity to read/write in English
* hospitalization in recent 6 months
* current drug or alcohol use disorder
* psychotic symptoms
* medical exclusion for use of NRT

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle R vanDellen, PhD, Principal Investigator — University of Georgia
Locations (1):
- University of Georgia, Athens, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with other researchers who request it.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Undecided
Access Criteria: Researchers must make request for data and materials to the PI

REFERENCES:
- [Derived] Andrade FC, Shen Y, MacKillop JM, Beach SRH, vanDellen MR. Dyadic patterns of abstinence from smoking in dual-smoking couples enrolled in a pilot randomized clinical trial. Health Psychol. 2026 Jan 29:10.1037/hea0001573. doi: 10.1037/hea0001573. Online ahead of print. PMID 41609650

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Dyad
Period: Overall Study
Arm/Group | Control (CTL) | Single Target (ST) | Dyadic Target (DT)
Started | 58; 29 Dyad | 68; 34 Dyad | 64; 32 Dyad
Completed | 54; 28 Dyad | 58; 30 Dyad | 58; 29 Dyad
Not Completed | 4; 1 Dyad | 10; 4 Dyad | 6; 3 Dyad

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control (CTL) | Single Target (ST) | Dyadic Target (DT) | Total
Number analyzed (Participants) | 58 | 68 | 64 | 190
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.67 (10.42) | 43 (10.90) | 42.4 (10.5) | 42.4 (10.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 35 | 34 | 99
  Male | 28 | 33 | 30 | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 9 | 4 | 15
  Not Hispanic or Latino | 36 | 39 | 40 | 115
  Unknown or Not Reported | 20 | 20 | 20 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 2
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 5 | 13 | 26
  White | 45 | 54 | 47 | 146
  More than one race | 2 | 3 | 2 | 7
  Unknown or Not Reported | 1 | 5 | 2 | 8
Region of Enrollment [Number; unit: participants]
  United States | 58 | 68 | 64 | 190
Education [Count of Participants; unit: Participants]
  Less than College Degree | 43 | 41 | 37 | 121
  College/Technical School Graduate | 14 | 23 | 21 | 58
  Post-college Education | 1 | 4 | 6 | 11
Relationship Length [Mean (Standard Deviation); unit: years] | 7.86 (8.48) | 7.44 (7.31) | 8.91 (8.65) | 8.06 (8.12)

OUTCOME MEASURES:

1. Primary Outcome: Smoking Abstinence
Description: Percentage of targets who have quit smoking by the follow-up study cessation verified biochemically
Time Frame: Follow-up study session 3 months post-baseline session
Measure: Number; unit: Targets
Units Other Than Participants: Targets
Arm/Group | Control (CTL) | Single Target (ST) | Dyadic Target (DT)
Number analyzed (Participants) | 58 | 68 | 64
Number analyzed (Targets) | 29 | 34 | 32
Targets
  Targets Abstinent | 4 | 16 | 9
  Targets Not Abstinent | 25 | 18 | 23

2. Primary Outcome: Feasibility of Financial Incentives Treatment in Dyadic-Smoker Couples
Description: Feasibility of financial incentives treatment in dyadic-smoker couples was assessed by number of individuals retained in study. Retention was separated by condition.
Time Frame: Through study recruitment and study completion, an average of five months
Measure: Count of Participants; unit: Participants
Arm/Group | Control (CTL) | Single Target (ST) | Dyadic Target (DT)
Number analyzed (Participants) | 58 | 68 | 64
Participants | 54 | 58 | 58

3. Primary Outcome: Tolerability of Financial Incentives Treatment in Dyadic-Smoker Couples
Description: Participant subjective ratings of the benefits and costs of participating in the study. Tolerability was defined using eight items assessing the accessibility, benefits, and costs of the study scored on a 1 (strongly disagree) to 7 (strongly agree) scale. Tolerability scores were separated by target and partner and reported by condition.
Time Frame: Through study recruitment and study completion, an average of five months
Population: Targets and Partners were analyzed separately. Thus, the total number of participants is 2x the number of targets and partners.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Control (CTL) | Single Target (ST) | Dyadic Target (DT)
Number analyzed (Participants) | 58 | 68 | 64
units on a scale
  Target Tolerability: number analyzed (Participants) | 29 | 34 | 32
  Target Tolerability | 4.99 [4.62 to 5.36] | 5.22 [4.95 to 5.49] | 4.99 [4.59 to 5.38]
  Partner Tolerability: number analyzed (Participants) | 29 | 34 | 32
  Partner Tolerability | 4.99 [4.67 to 5.32] | 5.04 [4.66 to 5.42] | 5.00 [4.60 to 5.40]

ADVERSE EVENTS:
Time Frame: Adverse events were collected during study participation (3 months)
Description: Adverse events were to be self-reported through email.
Arm/Group | Control (CTL) | Single Target (ST) | Dyadic Target (DT)
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/68 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/68 | 0/64
Other Adverse Events (participants affected / at risk) | 0/58 | 0/68 | 0/64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-21): https://cdn.clinicaltrials.gov/large-docs/60/NCT04832360/Prot_SAP_001.pdf
  • Informed Consent Form (2020-11-11): https://cdn.clinicaltrials.gov/large-docs/60/NCT04832360/ICF_000.pdf